CLINICAL TRIAL: NCT06189287
Title: Survey on Patients' Knowledge of Anesthesia Ethics and Research
Brief Title: Ethics and Research in Anaesthesia
Acronym: Anesth_ethic
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB_23.03.09
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Ethics, Narrative; Surgery
MeSH Terms: conditions — Narration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patient of legal age agreeing to answer an anonymous questionnaire on their knowledge of clinical research given at the anesthesia consultation for scheduled surgery

SUMMARY:
Under the impetus of governing bodies, learned societies, hospital management, CPPs, etc., clinical research has developed and structured considerably, in order to provide the medical community and patients with the most appropriate care, and to formulate recommendations.

In anesthesia, clinical research evaluates drugs, medical devices or care pathways. However, the general public's perception of this research in our specialty remains confidential. Several studies carried out in oncology have shown limited interest in research on the part of the general public and patients, and more often than not a lack of awareness of ethical laws and the role of french ethics committee (CPP).

By means of an anonymous questionnaire handed out at the anesthesia consultation, the investigators would like to assess patients' level of knowledge of clinical research in anesthesia, and find out how they feel about the possibility of being included in a trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* patient undergoing surgery

Exclusion Criteria

* Refusal to participate
* Patient unable to read or answer questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients over 18 years of age scheduled for surgery who agree to answer the survey
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Survey response | Day 0
  descriptive data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Principal Investigator — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No